CLINICAL TRIAL: NCT05284435
Title: Internet-Based, Parent-Led Cognitive-Behavioral Therapy for Anxiety in Youth With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Andrew Guzick, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-51359
Record Dates: First submitted 2022-03-09; First posted 2022-03-17 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Cognitive Behavioral Therapy; Autism Spectrum Disorder; Anxiety Disorder; Obsessive-Compulsive Disorder; Social Anxiety Disorder; Generalized Anxiety Disorder; Specific Phobia
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Obsessive-Compulsive Disorder; Phobia, Social; Generalized Anxiety Disorder; Phobia, Specific

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCBT-Email (iCBT-E) (Experimental): Parents will receive a weekly email from a therapist over the 12 weeks of treatment.
  Interventions: Behavioral: Cognitive Behavioral Therapy-Email (iCBT-E)
- iCBT-Email and Videoconferencing (iCBT-EV) (Active Comparator): Parents will receive a weekly email and six 30-minute supportive video calls with a therapist over the 12 weeks of treatment.
  Interventions: Behavioral: Cognitive Behavioral Therapy-Email and Videoconferencing (iCBT-EV)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy-Email (iCBT-E) — Participating families will receive an access to the website that contains treatment materials for both parent and child.
  During each of the weekly emails, therapists will serve to provide encouragement and support as the parent works through the program independently.
  Arms: iCBT-Email (iCBT-E)
Behavioral: Cognitive Behavioral Therapy-Email and Videoconferencing (iCBT-EV) — Participating families will receive an access to the website that contains treatment materials for both parent and child.
  During each of the weekly emails and six videoconferencing sessions, therapists will serve to provide encouragement and support as the parent works through the program independently. Therapists will also assist the parent with any problem-solving as needed.
  Arms: iCBT-Email and Videoconferencing (iCBT-EV)

SUMMARY:
This study compares the effectiveness of two levels of therapist support for an internet-based, parent-led cognitive behavioral therapy for youth with anxiety and ASD.

DETAILED DESCRIPTION:
Autism spectrum disorder, or ASD, is one of the most common neurodevelopmental disorders, affecting up to 1 out of 59 youth in the United States. Anxiety disorders affect 50-80% of children with ASD and are associated with significant life impairment and worsening trajectory without treatment. Cognitive-behavioral therapy (CBT) is an effective treatment for anxiety, yet access to CBT is very limited for most families due to the cost, practicalities of attending in-person treatment sessions and limited availability of trained therapists. Access to CBT is particularly limited for Hispanic or Spanish-speaking families due to lack of services provided in Spanish. Web-based or internet-based delivery of services is a promising method to improve access to care for youth with ASD and their families, given its reachability to a wider range of areas (e.g., rural/underserved) and its ability to minimize practical barriers (e.g., treatment could be delivered to home without need for travel), and reduce stigma (e.g., parents do not need to visit mental health clinics). Thus, the goal of this project is to increase access to care for families of children with ASD and anxiety through an internet-based treatment intervention model. This intervention, developed by the study team, consists of an interactive website with treatment materials that parents can work through with their child, both in English and Spanish.

Specifically, this project will examine the effectiveness of an internet-based, parent-led cognitive-behavioral therapy (iCBT) for anxiety in children with two levels of therapist support: 1) iCBT-E (therapist support is delivered via email) and 2) iCBT-EV (therapist support is delivered via email and videoconferencing sessions).

This study will also involve two phases: 1) pilot intervention phase and 2) randomized controlled phase.

ELIGIBILITY:
Inclusion Criteria:

* Child is between the ages 7-15 years at consent/assent.
* The child meets criteria for ASD.
* The child meets criteria for an anxiety and/or obsessive compulsive disorder (OCD) as determined by the Mini Neuropsychiatric Interview for Children and Adolescents
* Anxiety and/or OCD is the primary presenting problem as determined by the Mini Neuropsychiatric Interview for Children and Adolescents
* One parent/guardian is able and willing to participate.
* The child has a Full Scale and Verbal Comprehension Intelligence Quotient >70.
* The child is able to communicate verbally.
* Participants must reside in Texas and must be in the state of Texas when taking calls.

Exclusion Criteria:

* The child has a diagnosis of lifetime DSM-5 bipolar disorder, psychotic disorder, and/or intellectual disability.
* The child has severe current suicidal/homicidal ideation and/or self-injury requiring medical intervention.
* The child is receiving concurrent psychotherapy for anxiety.
* Initiation of a psychotropic medication less than 4 weeks prior to study enrollment or a stimulant/psychoactive medication less than 2 weeks prior to study enrollment.

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-12-17 (Actual)

PRIMARY OUTCOMES:
5-item Pediatric Anxiety Rating Scale - Autism Spectrum Disorder | 7 days
  Clinician rated child anxiety severity throughout the past week. Each item is scored on a 0 to 5 scale (higher scores correspond to greater severity), yielding a total between 0 and 30.
Clinical Global Impression-Improvement | 7 days
  Clinician rated child psychopathology improvement since initial rating. A single item is scored 0-6 (0 = very much worse; 6= very much improved).

SECONDARY OUTCOMES:
Revised Child Anxiety and Depression Scale- Parent-Report- Anxiety Subscale | 7 days
  Parent rated child anxiety severity. It is a 37-item scale and each item is scored on a 0 ("never") to 3 ("always") scale (higher scores correspond to greater severity), yielding a total between 0 to 111.
Revised Child Anxiety and Depression Scale- Self-Report- Anxiety Subscale | 7 days
  Child rated anxiety severity. It is a 37-item scale and each item is scored on a 0 ("never") to 3 ("always") scale (higher scores correspond to greater severity), yielding a total between 0 to 111.
Social Responsiveness Scale, Second Edition | 7 days
  Parent rated child impairment in social behaviors. It is a 65-item scale and each item is scored on a 1 ("not true") to 4 ("almost always true") scale (higher scores correspond to greater impairment), yielding a total raw score between 65 and 260.
Sheehan Disability Scale | 7 days
  Parent rated child functional impairment. It is a 5-item scale and each item is scored on a 0 ("not at all") to 10 ("extremely") scale (higher scores correspond to greater impairment), yielding a total between 0 and 50.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guzick AG, Schneider SC, Kook M, Greenberg R, Perozo-Garcia A, Lee MP, Garcia J, Onyeka OC, Riddle DB, Storch EA. Internet-based, parent-led cognitive behavioral therapy for autistic youth with anxiety-related disorders: A randomized trial comparing email vs. telehealth support. Behav Res Ther. 2024 Dec;183:104639. doi: 10.1016/j.brat.2024.104639. Epub 2024 Sep 29. PMID 39368459